CLINICAL TRIAL: NCT02126449
Title: DIetary REstriction as an Adjunct to Neoadjuvant ChemoTherapy for HER2 Negative Breast Cancer
Acronym: DIRECT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Borstkanker Onderzoek Groep (Network); Pink Ribbon Inc. (Industry); Amgen (Industry)
Responsible Party: Principal Investigator, J.R. Kroep, MD, PhD, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL44684.058.13; BOOG2013-04 (Other: BOOG); p13.135 (Other: CME LUMC)
Record Dates: First submitted 2014-02-14; First posted 2014-04-30 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Fasting Mimicking Diet; Breast Cancer; Neoadjuvant Chemotherapy; Pathological Complete Response
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fasting mimicking diet (Experimental): Short term fasting using Fasting mimicking diet around neoadjuvant chemotherapy (AC>T)
  Interventions: Other: Fasting mimicking diet
- regular diet (No Intervention): Standard neoadjuvant chemotherapy (AC>T)

INTERVENTIONS:
Other: Fasting mimicking diet
  Arms: Fasting mimicking diet

SUMMARY:
Preclinical studies provide strong support for the concept that fasting evokes resistance to multiple forms of stress. Fasting reduces plasma levels of growth factors and modulates intracellular nutrient sensing systems, thereby diverting energy from growth to maintenance. Accordingly, the currently available preclinical evidence suggests that short-term fasting protects normal cells against the perils of chemotherapy. In contrast, cancer cells are not protected, as a result of their self-sufficiency in growth signals. This phenomenon is termed Differential Stress Resistance (DSR). DSR reduces the severity of toxic side-effects of chemotherapy and interestingly, it simultaneously renders cancer cells more vulnerable to chemotherapeutics. Importantly, extensive preclinical evidence and preliminary clinical data indicate that a specifically designed very low calorie, low amino acid substitution diet ("Fasting Mimicking Diet, FMD") has effects on cancer therapy that are very similar to those of fasting. This study aims to evaluate the impact of the FMD on tolerance to and efficacy of neoadjuvant chemotherapy in women with stage II or III breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with stage II or III (cT1cN+ or ≥T2 any cN, cM0) breast cancer receiving neoadjuvant AC-T
* Measurable disease (breast and/or lymph nodes)
* HER2 negative core biopsy Age ≥18 years
* WHO performance status 0-2
* Adequate bone marrow function : white blood cells (WBCs) ≥3.0 x 109/l, neutrophils ≥1.5 x 109/l, platelets ≥100 x 109/l
* Adequate liver function: bilirubin ≤1.5 x upper limit of normal (UNL) range, ALAT and/or ASAT ≤2.5 x UNL, Alkaline Phosphatase ≤5 x UNL
* Adequate renal function: the calculated creatinine clearance should be ≥50 mL/min
* Patients must be accessible for treatment and follow-up
* Written informed consent according to the local Ethics Committee requirements
* Willing to fill in quality of life questionnaires
* Able to read and write in Dutch

Exclusion Criteria:

* History of breast cancer (invasive or non-invasive)
* Previous malignancy within 5 years, with exception of a history of a previous basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix.
* Serious other diseases such as recent myocardial infarction, clinical signs of cardiac failure or clinically significant arrhythmias
* Diabetes Mellitus
* Body mass index (BMI) < 19 kg/m2
* Pregnancy or lactating
* Significant food allergies which would make the subject unable to consume the food provided (ex: nuts or soy)
* Any metabolic disorders that may affect gluconeogenesis or adaptation to short fasting periods.
* Medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or sign meaningful informed consent

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
The percentage of patients with grade III/IV toxicity according to the National Cancer Institute Common Terminology Criteria for Adverse Events version (NCI CTCAE) v4.03. | 2 years
  Phase II
The percentage of pCR. | 4 years
  Phase III

SECONDARY OUTCOMES:
Clinical response measured by MRI (RECIST1.1) after 4 cycles chemotherapy. | 4 years
Grade I/II side effects of chemotherapy according to NCI CTCAE v4.03. | 4 years
Metabolic (Glucose, insulin, insulin-like growth factor-I (IGF-I), insulin-like growth factor binding protein 3 (IGF-BP3), free thyroxin (FT4), triiodothyronine (T3) and thyroid-stimulating hormone (TSH)) and inflammatory response (CRP) to chemotherapy. | 4 years
DNA damage, apoptosis, immunology and nutrient sensing system activity in the tumor. | 5 years
Patient's quality of life (using EORTC QLQ-C30 and EORTC QLQ-BR23 questionnaires), burden of therapy noted by a visual analogue scale (VAS) (Distress Thermometer) and differences of Illness Perceptions (B-IPQ). | 4 years
Long term efficacy of treatment (DFS, OS). | 4years
Hormone receptor percentage, Ki67 and immunologic tumor profile and tumor/stroma ratio as predictive biomarker | 4 years
SNPs used as biomarker to predict treatment outcome. | 5 years

OTHER OUTCOMES:
Protein profiles and cytokines used as biomarker to predict treatment outcome | 4 years
Quantification of chemotherapy-induced DNA damage in leukocytes (with γ-H2AX modification and comet assay). | 3years
Quantification of nutrient sensing system gene expression (with western blot). | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Judith R Kroep, MD, PhD, Principal Investigator — Leiden University Medical Center; Hanno Pijl, MD PhD, Principal Investigator — Leiden University Medical Center; Koos JM van der Hoeven, MD PhD Ir, Principal Investigator — Leiden University Medical Center
Locations (15):
- Netherlands (15):
  - Leids Universitair Medisch Centrum, Leiden, South Holland
  - Medisch Centrum Alkmaar, Alkmaar
  - OLVG, Amsterdam
  - Alexander Monro hospital, Bilthoven
  - Amphia Hospital, Breda
  - Deventer Hospital, Deventer
  - Ziekenhuis Gelderse Valei, Ede
  - , Catharina ziekenhuis Hospital, Eindhoven
  - Kennemer gasthuis, Haarlem
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Bronovo Hospital, The Hague
  - Haga Hospital, The Hague
  - VieCurie Hospital, Venlo
  - Lange Land Hospital, Zoetermeer
  - Isala, Zwolle

REFERENCES:
- [Derived] Lugtenberg RT, de Groot S, Kaptein AA, Fischer MJ, Kranenbarg EM, Carpentier MD, Cohen D, de Graaf H, Heijns JB, Portielje JEA, van de Wouw AJ, Imholz ALT, Kessels LW, Vrijaldenhoven S, Baars A, Fiocco M, van der Hoeven JJM, Gelderblom H, Longo VD, Pijl H, Kroep JR; Dutch Breast Cancer Research Group (BOOG). Quality of life and illness perceptions in patients with breast cancer using a fasting mimicking diet as an adjunct to neoadjuvant chemotherapy in the phase 2 DIRECT (BOOG 2013-14) trial. Breast Cancer Res Treat. 2021 Feb;185(3):741-758. doi: 10.1007/s10549-020-05991-x. Epub 2020 Nov 11. PMID 33179154
- [Derived] de Groot S, Lugtenberg RT, Cohen D, Welters MJP, Ehsan I, Vreeswijk MPG, Smit VTHBM, de Graaf H, Heijns JB, Portielje JEA, van de Wouw AJ, Imholz ALT, Kessels LW, Vrijaldenhoven S, Baars A, Kranenbarg EM, Carpentier MD, Putter H, van der Hoeven JJM, Nortier JWR, Longo VD, Pijl H, Kroep JR; Dutch Breast Cancer Research Group (BOOG). Fasting mimicking diet as an adjunct to neoadjuvant chemotherapy for breast cancer in the multicentre randomized phase 2 DIRECT trial. Nat Commun. 2020 Jun 23;11(1):3083. doi: 10.1038/s41467-020-16138-3. PMID 32576828
- See also: Related Info — https://www.boogstudycenter.nl